CLINICAL TRIAL: NCT02877680
Title: Development and Pilot of a Strengths-Based Behavioral mHealth Intervention to Promote Resilience in Adolescents With Type 1 Diabetes
Brief Title: Strengths-Based Behavioral mHealth App for Parents of Adolescents With Type 1 Diabetes-Pilot Study
Acronym: T1DoingWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northwestern University Feinberg School of Medicine (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marisa Hilliard, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37311; 1R21DK107951 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Strengths-based; Mobile Health (mHealth); Adolescence; Resilience; Family
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Smartphone app for parents to track adolescents' strength behaviors related to living with and managing type 1 diabetes, including regular feedback to parents and training about how to recognize and reinforce positive behaviors in teens.
  Interventions: Behavioral: T1Doing Well
- Usual Care (No Intervention): Usual diabetes care and study-related data collection, without use of app during the study period. They will be offered an opportunity to try the app and share their feedback with the study team after completing follow-up data collection.

INTERVENTIONS:
Behavioral: T1Doing Well — Strengths-based mobile health (mHealth) app for parents of adolescents with type 1 diabetes, which will prompt parents to recognize and reinforce their adolescents' diabetes-related strength behaviors
  Arms: Intervention

SUMMARY:
Type 1 diabetes (T1D) management is particularly challenging during adolescence as responsibility for management begins to shift from parents to youth, and positive family teamwork is critical to achieving optimal diabetes outcomes. Existing behavioral family interventions for T1D are beneficial but have limited potential for translation to clinical practice, and universal preventive approaches designed to explicitly promote existing T1D management strengths are needed. Ultimately, the goal of this line of research is to validate brief, convenient, and helpful tools that families of all adolescents with T1D can use to strengthen positive family teamwork and ultimately promote optimal diabetes health outcomes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is among the most common chronic conditions of childhood and its management is complex and relentless. Adolescents have increased risk for worsening glycemic control, putting them at risk for short- and long-term complications. As responsibility for daily T1D management tasks begins to shift from parents to youth, supportive parent-adolescent teamwork promotes optimal diabetes outcomes. However, adolescents' cognitive development, desire for autonomy, and changing family and social relationships can make adherence to treatment recommendations difficult and strain attempts at parent-adolescent teamwork. This study aims to develop and pilot test a mobile app-based behavioral intervention to facilitate positive, supportive parent-adolescent interactions around T1D management. The proposed study has two parts. First, adolescents with T1D (age 12-17), their parents, and diabetes care providers will be invited to participate in designing a smartphone app that supports parents to recognize, keep track of, and reinforce their adolescents for specific positive T1D-related behaviors, or strengths. Example strengths include asking for help with complicated diabetes tasks, talking to friends about diabetes, and expressing confidence or optimism about T1D management. Intermittently throughout the day, the app will push parents a prompt to report which positive T1D behaviors their adolescent has engaged in. The app will generate weekly summary reports of each adolescent's most frequent strength behaviors, and parents will be reminded via the app to praise their adolescent for those patterns. Second, this intervention will be pilot tested with 82 families; parents will be randomized to an intervention or a control condition. Participants in the intervention condition will use the app for 3-4 months and provide feedback, and control participants will receive usual care and will not use the app. The main goal is to determine how often and in what ways families use the app, whether they like it, and to obtain suggestions for improvement. Trends for impact on important diabetes outcomes, such as quality of parent-adolescent relationships, T1D treatment adherence, and glycemic control will also be evaluated. Data - including questionnaires, adherence data from blood glucose meters, and glycemic control biomarkers from a blood draw - will be collected at baseline and again 3-4 months later. The results of this pilot study will help refine the intervention so that it can be evaluated in a fullscale randomized controlled trial. Ultimately, the goal of this research is to validate brief, convenient, and helpful tools that families of all adolescents with T1D can use to strengthen positive family teamwork and ultimately promote optimal diabetes health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes according to American Diabetes Association criteria for at least 6 months
* Treated for type 1 diabetes at Texas Children's Hospital Diabetes Care Center
* Parent and adolescent fluency in English
* Parent has mobile device with data plan

Exclusion Criteria:

* Serious medical, cognitive, or mental health comorbidity in parent or adolescent that would preclude ability to participate

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa E Hilliard, PhD, Principal Investigator — Baylor College of Medicine and Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual health data will be collected that is not already available to families through their electronic medical record

REFERENCES:
- [Derived] Hilliard ME, Cao VT, Eshtehardi SS, Minard CG, Saber R, Thompson D, Karaviti LP, Anderson BJ. Type 1 Doing Well: Pilot Feasibility and Acceptability Study of a Strengths-Based mHealth App for Parents of Adolescents with Type 1 Diabetes. Diabetes Technol Ther. 2020 Nov;22(11):835-845. doi: 10.1089/dia.2020.0048. Epub 2020 May 22. PMID 32379496
- [Derived] Hilliard ME, Eshtehardi SS, Minard CG, Saber R, Thompson D, Karaviti LP, Rojas Y, Anderson BJ. Strengths-Based Behavioral Intervention for Parents of Adolescents With Type 1 Diabetes Using an mHealth App (Type 1 Doing Well): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2018 Mar 13;7(3):e77. doi: 10.2196/resprot.9147. PMID 29535081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from diabetes clinics at Texas Children's Hospital.
Pre-assignment Details: Of 84 families consented, 2 families did not complete baseline questionnaires and were not randomized (1 withdrew due to time demands, 1 moved to another care institution). Of the remaining 82 families, 2 completed baseline questionnaires but were never randomized because they never completed a study visit, resulting in a randomized sample of n=80.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 55 | 25
Completed | 54 | 24
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of 84 families (parent-adolescent dyads) consented, n=4 were never randomized (reasons stated in Participant Flow section), resulting in baseline data from 80 families.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 55 | 25 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.5) | 15.1 (1.4) | 15.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Adolescent: Female | 33 | 14 | 47
  Adolescent: Male | 22 | 11 | 33
  Parent: Female | 44 | 21 | 65
  Parent: Male | 11 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: Hispanic or Latino | 14 | 1 | 15
  Adolescent: Not Hispanic or Latino | 41 | 24 | 65
  Adolescent: Unknown or Not Reported | 0 | 0 | 0
  Parent: Hispanic or Latino | 14 | 1 | 15
  Parent: Not Hispanic or Latino | 40 | 24 | 64
  Parent: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: American Indian or Alaska Native | 0 | 0 | 0
  Adolescent: Asian | 1 | 0 | 1
  Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Adolescent: Black or African American | 8 | 2 | 10
  Adolescent: White | 39 | 20 | 59
  Adolescent: More than one race | 4 | 3 | 7
  Adolescent: Unknown or Not Reported | 3 | 0 | 3
  Parent: American Indian or Alaska Native | 0 | 0 | 0
  Parent: Asian | 1 | 0 | 1
  Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Parent: Black or African American | 8 | 2 | 10
  Parent: White | 41 | 21 | 62
  Parent: More than one race | 0 | 2 | 2
  Parent: Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 55 | 25 | 80
Adherence to Diabetes Regimen (Objective) - Blood Glucose Monitoring Frequency [Mean (Standard Deviation); unit: Checks per day] — Objective measurement of adherence to diabetes regimen measured by blood glucose monitoring frequency (a well-accepted surrogate of overall adherence), obtained via blood glucose meter downloads. The average daily frequency was calculated over the 14 days prior to the assessment at the baseline visit. Population: n represents number with complete data.
  Checks per day
    number analyzed (Participants) | 51 | 22 | 73
    (all) | 2.9 (1.8) | 3.2 (1.4) | 3.0 (1.7)
Glycemic control - HbA1c [Mean (Standard Deviation); unit: percentage] — At the time of this study, the American Diabetes Association generally recommended an HbA1c target of <7.5% for individuals younger than 18 years (specific target varies depending on the individual). The DCA 2000 HbA1c Analyzer (Siemens-Bayer) was used for point of care HbA1c analysis, it has an analytical measurement range for HbA1c of 2.5% to 14.0%. HbA1c values are collected via fingerstick and blood assay at routine diabetes care visits and values were extracted from the medical record at each clinic visit during the study period. Population: n is the number with an HbA1c value available at this timepoint.
  percentage
    number analyzed (Participants) | 55 | 24 | 79
    (all) | 9.1 (2.1) | 8.7 (2.1) | 9.0 (2.1)
Diabetes Family Impact - Diabetes Family Impact Scale (DFIS), Parent-report [Mean (Standard Deviation); unit: units on a scale] — Diabetes-specific family impact was measured using the Diabetes Family Impact Scale (DFIS), a 15-item measure of the impact of diabetes on family members' activities and relationships. The scale range from the minimum to maximum possible score is 0-100. A higher score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 54 | 25 | 79
    (all) | 20.0 (12.9) | 20.3 (17.7) | 20.12 (14.5)
Family Impact - Pediatric Quality of Life Family Impact Module (Peds QL-FI), Parent-report [Mean (Standard Deviation); unit: units on a scale] — Family impact was measured using the Diabetes Family Impact Scale (DFIS), a 15-item measure of the impact of diabetes on family members' activities and relationships. The scale ranges from 0-100. A higher score represents a better outcome.
  units on a scale | 83.7 (13.6) | 83.9 (13.2) | 83.8 (13.4)
Family Communication - Helping for Health Inventory (HHI), Parent report [Mean (Standard Deviation); unit: units on a scale] — Family communication was measured by the parent-report Helping for Health Inventory (HHI), a 15-item measure of perceptions of parental help around the teen's diabetes management. The scale range from the minimum to maximum possible score is 15-75. A lower score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 51 | 24 | 75
    (all) | 39.6 (11.0) | 39.0 (9.2) | 39.4 (10.4)
Family Communication - Helping for Health Inventory (HHI), Adolescent report [Mean (Standard Deviation); unit: units on a scale] — Family communication was measured with the Helping for Health Inventory (HHI), a 15-item measure of perceptions of parental help around the teen's diabetes management. The scale range from the minimum to maximum possible score is 15-75. A lower score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 55 | 23 | 78
    (all) | 40.1 (11.6) | 41.4 (12.0) | 40.5 (11.7)
Diabetes Family Conflict Scale-Revised (DCFS), Parent-report [Mean (Standard Deviation); unit: units on a scale] — Family conflict was measured using the Diabetes Family Conflict Scale - Revised (DFCS), a measure of diabetes-specific conflict in families with adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 19-57. A lower score represents a better outcome.
  units on a scale | 26.7 (6.1) | 25.2 (3.5) | 26.2 (5.5)
Diabetes Family Conflict Scale-Revised (DFCS), Adolescent-report [Mean (Standard Deviation); unit: units on a scale] — Family conflict was measured using the Diabetes Family Conflict Scale-Revised (DFCS), a measure of diabetes-specific conflict in families with adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 19-57. A lower score represents a better outcome.
  units on a scale | 24.5 (4.7) | 26.5 (8.4) | 25.1 (6.1)
Problem Areas in Diabetes-Teen (PAID-T), Parent-report [Mean (Standard Deviation); unit: units on a scale] — Diabetes burden was measured using the Problem Areas in Diabetes (PAID-T) parent-report, a measure of how bothersome day-to-day problems are for parents of adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 26-156. A lower score represent better a outcome.
  units on a scale | 73.9 (21.9) | 68.4 (18.9) | 72.2 (21.0)
Problem Areas in Diabetes-Teen (PAID-T), Adolescent Self-report [Mean (Standard Deviation); unit: units on a scale] — Diabetes burden was measured using the Problem Areas in Diabetes-Teen (PAID-T) self-report, a measure of how bothersome day-to-day problems are for adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 26-156. A lower score represents better a outcome.
  units on a scale | 63.5 (25.8) | 63.5 (29.8) | 63.5 (26.9)
Self-Management - Diabetes Self-Management Profile (DSMP), Parent-report [Mean (Standard Deviation); unit: units on a scale] — Parent report of adolescent's self-management was measured using the 24-item Diabetes Self-Management Profile Self-Report (DSMP). The version appropriate to their child's current diabetes regimen (conventional insulin regimen, 24 items; flexible insulin regimen, 24 items) was administered. The scale range from the minimum to maximum possible score is 0-86. A higher score represents a better outcome.
  units on a scale | 52.1 (12.8) | 52.3 (10.5) | 52.1 (12.1)
Self-Management - Diabetes Self-Management Profile (DSMP), Adolescent Self-report [Mean (Standard Deviation); unit: units on a scale] — Parent-report of adolescent self-management was measured using the 24-item Diabetes Self-Management Profile Self-Report (DSMP). Parents completed the version appropriate to their child's current diabetes regimen (conventional insulin regimen, 24 items; flexible insulin regimen, 24 items). The scale range from the minimum to maximum possible score is 0-86. A higher score represents a better outcome.
  units on a scale | 69.1 (13.2) | 66.3 (15.1) | 68.2 (13.8)
Diabetes Strengths and Resilience Measure (DSTAR), Adolescent Self-report [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Strengths and Resilience (DSTAR) measure is a self-report assessment of positive behaviors related to diabetes resilience for youth with type 1 diabetes, such as perceived competence to manage the demanding diabetes regimen, to adapt to the unpredictability of diabetes, and to seek help and support with diabetes challenges. The scale range from the minimum to maximum possible score is 0-48. A higher score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 53 | 25 | 78
    (all) | 37.6 (6.3) | 34.8 (5.3) | 36.7 (6.1)
Adolescent Quality of Life - The MIND-Youth Questionnaire, Adolescent self-report [Mean (Standard Deviation); unit: units on a scale] — Adolescent quality of life was measured using the Monitoring Individual Needs in Diabetes Youth Questionnaire (MIND-Youth/MY-Q), a 33-item measure of diabetes-specific health-related QOL. The scale range from the minimum to maximum possible score is 0-100. A higher score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 54 | 25 | 79
    (all) | 72.3 (12.9) | 70.7 (15.1) | 71.8 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Design - Recruitment Rate
Description: Recruitment data measured by percent of recruited families that enrolled in study.
Time Frame: Immediately following enrollment (baseline timepoint)
Population: Out of 108 families successfully contacted and confirmed eligible, 8 families declined due to time demands, 6 were disinterested in research, and 2 felt the study was not relevant for their child's age. 8 families were unable to be contacted for a decision after giving study information. 84 families consented (78% consent rate).
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent-Parent Dyads: Upon recruitment and enrollment, families completed baseline questionnaires. After baseline questionnaire completion, families were randomized 2:1 to (A) intervention group where parents use a strengths-based mobile health (mHealth) app, which will prompt parents to recognize and reinforce their adolescents' diabetes-related strength behaviors, or (B) usual diabetes care group, without use of app during the study period.
  Both groups completed the same follow-up surveys. Additionally, intervention parents completed a set of follow-up questionnaires about usability of the app, and intervention families were asked to participate in an exit interview to share their experiences with the app.
Arm/Group | Adolescent-Parent Dyads
Number analyzed (Participants) | 108
Participants | 84

2. Primary Outcome: Feasibility of T1Doing Well App - Engagement With App At Least Twice A Week
Description: Feasibility of the app measured by percentage of participants that engaged with or used the app at least twice a week during the intervention period.
Time Frame: 3-4 months after enrollment (follow-up timepoint)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 55
Participants | 50

3. Primary Outcome: Acceptability of T1Doing Well App (Survey)
Description: Participants in the intervention arm completed the Usefulness, Satisfaction, and Ease of Use Questionnaire (USE), a measure of the users' perceived usefulness of, satisfaction with, and ease of use of a particular technology. The item scale ranges from the minimum to maximum possible score is 1-7, with a higher score representing a better outcome. Acceptability measured as percentage of participants who selected a score of at least 4 (out of 7) on the item "I am satisfied with it," indicating it was at least somewhat acceptable.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 55
Participants | 48

4. Primary Outcome: Acceptability - Number of Participants That Felt The Intervention Was Well-Received
Description: The number of participants that felt the intervention was well-received was collected for Adolescents and Parents. To determine if the intervention was well-received, verbal responses from qualitative interviews with were coded for types of participant feedback by the study team. We coded these data qualitatively and classified them as Positive, Negative, or Neutral. Positive responses indicate the intervention was well-received.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number we were able to reach and obtain follow-up interview data
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Parent; Intervention - Adolescent: Smartphone app for parents to track adolescents' strength behaviors related to living with and managing type 1 diabetes, including regular feedback to parents and training about how to recognize and reinforce positive behaviors in teens.
  T1Doing Well: Strengths-based mobile health (mHealth) app for parents of adolescents with type 1 diabetes, which will prompt parents to recognize and reinforce their adolescents' diabetes-related strength behaviors.
Arm/Group | Intervention - Parent | Intervention - Adolescent
Number analyzed (Participants) | 46 | 47
Participants | 35 | 38

5. Secondary Outcome: Adherence to Diabetes Regimen (Objective) - Blood Glucose Monitoring Frequency
Description: Objective measurement of adherence to diabetes regimen measured by blood glucose monitoring frequency (a well-accepted surrogate of overall adherence), obtained via blood glucose meter downloads. The average daily frequency was calculated over the 14 days prior to the assessment at the baseline visit.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: Checks per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 33 | 18
Checks per day | 2.6 (1.9) | 3.1 (1.2)

6. Secondary Outcome: Glycemic Control - HbA1c
Description: At the time of this study, the American Diabetes Association generally recommended an HbA1c target of <7.0% (it was <7.5% at the time this study took place, for individuals younger than 18 years. The especific target varies depending on the individual). The DCA 2000 HbA1c Analyzer (Siemens-Bayer) was used for point of care HbA1c analysis, it has an analytical measurement range for HbA1c of 2.5% to 14.0%. HbA1c values are collected via fingerstick and blood assay at routine diabetes care visits and values were extracted from the medical record at each clinic visit during the study period.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n is the number with an HbA1c value available at this timepoint.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 51 | 22
percentage | 8.7 (1.7) | 8.4 (1.4)

7. Secondary Outcome: Diabetes Family Impact - Diabetes Family Impact Scale (DFIS), Parent-report
Description: Diabetes-specific family impact was measured using the Diabetes Family Impact Scale (DFIS), a 15-item measure of the impact of diabetes on family members' activities and relationships. The scale range from the minimum to maximum possible score is 0-100. A higher score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 24
units on a scale | 20.7 (15.5) | 19.1 (16.1)

8. Secondary Outcome: Family Impact - Pediatric Quality of Life Impact Module (Peds QL-FI), Parent-report
Description: Family impact was measured using The Pediatric Quality of Life Family Impact Module (Peds QL-FI), a 36-item measure of the impact of parenting a child with a chronic medical condition on family functioning and parent QOL. The scale range from the minimum to the maximum score is 0-100. A higher score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 24
units on a scale | 82.6 (14.1) | 84.5 (15.4)

9. Secondary Outcome: Family Communication - Helping for Health Inventory (HHI), Parent-report
Description: Family communication was measured by the parent-report Helping for Health Inventory (HHI), a 15-item questionnaire assessing perceptions of parental help around the teen's diabetes management. The scale range from the minimum to maximum possible score is 15-75. A lower score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 52 | 24
units on a scale | 40.0 (12.5) | 40.0 (9.9)

10. Secondary Outcome: Family Communication - Helping for Health Inventory (HHI), Adolescent-report
Description: Family communication was measured using the adolescent-report Helping for Health Inventory (HHI), a 15-item questionnaire assessing perceptions of parental help around the teen's diabetes management. The scale range from the minimum to maximum possible score is 15-75. A lower score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 51 | 23
units on a scale | 37.9 (10.6) | 41.4 (13.1)

11. Secondary Outcome: Diabetes Family Conflict Scale-Revised (DFCS), Parent-report
Description: Family conflict was measured using the Diabetes Family Conflict Scale - Revised (DFCS), a measure of diabetes-specific conflict in families with adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 19-57. A lower score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 24
units on a scale | 25.4 (5.2) | 24.5 (3.9)

12. Secondary Outcome: Diabetes Family Conflict Scale-Revised (DFCS), Adolescent-report
Description: as for outcome 11
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 24
units on a scale | 23.9 (4.5) | 25.0 (6.2)

13. Secondary Outcome: Problem Areas in Diabetes-Teen (PAID-T), Parent-report
Description: Diabetes burden was measured using the Problem Areas in Diabetes (PAID-T) parent-report, a measure of how bothersome day-to-day problems are for parents of adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 26-156. A lower score represents better a outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 55 | 24
units on a scale | 77.6 (28.1) | 71.0 (28.4)

14. Secondary Outcome: Problem Areas in Diabetes-Teen (PAID-T), Adolescent Self-report
Description: Diabetes burden was measured using the Problem Areas in Diabetes-Teen (PAID-T) self-report, a measure of how bothersome day-to-day problems are for adolescents with type 1 diabetes. The scale range from the minimum to maximum possible score is 26-156. A lower score represents better a outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 53 | 24
units on a scale | 65.0 (26.1) | 65.2 (25.7)

15. Secondary Outcome: Self-Management - Diabetes Self-Management Profile (DSMP), Parent-report
Description: Parent-report of adolescent self-management was measured using the 24-item Diabetes Self-Management Profile Self-Report (DSMP). Parents completed the version appropriate to their child's current diabetes regimen (conventional insulin regimen, 24 items; flexible insulin regimen, 24 items). The scale range from the minimum to maximum possible score is 0-86. A higher score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 24
units on a scale | 53.4 (10.8) | 53.0 (9.6)

16. Secondary Outcome: Self-Management - Diabetes Self-Management Profile (DSMP), Adolescent Self-report
Description: Self-management was measured using the Self-Care Inventory-Revised (SCI-R), a 15-item measure of the frequency that adolescents engage in diabetes management behaviors on a 5-point scale from Never to Always. The scale range from the minimum to maximum possible score is 5-75. A higher score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 54 | 25
units on a scale | 66.6 (14.0) | 68.4 (12.9)

17. Secondary Outcome: Diabetes Strengths and Resilience Measure (DSTAR), Adolescent Self-report
Description: The Diabetes Strengths and Resilience measure is a self-report assessment of positive behaviors related to diabetes resilience for youth with type 1 diabetes, such as perceived competence to manage the demanding diabetes regimen, to adapt to the unpredictability of diabetes, and to seek help and support with diabetes challenges. The scale range from the minimum to maximum possible score is 0-48. A higher value on this scale represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 52 | 25
units on a scale | 37.7 (5.7) | 35.1 (5.6)

18. Secondary Outcome: Adolescent Quality of Life - The MIND-Youth Questionnaire, Adolescent Self-report
Description: Adolescent quality of life was measured using the Monitoring Individual Needs in Diabetes Youth Questionnaire (MIND-Youth/MY-Q), a 33-item measure of diabetes-specific health-related QOL. The scale range from the minimum to maximum possible score is 0-100. A higher score represents a better outcome.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Population: n represents number with complete data to calculate a score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 53 | 24
units on a scale | 72.2 (11.8) | 68.4 (13.8)

19. Secondary Outcome: Parent-Adolescent Relationship Intervention Process Measure, Adolescent Report
Description: Adolescents answered 3 items adapted from the Parent-Youth Relationship Index of the National Longitudinal Study of Youth-1997, a measure of parent-adolescent relationship quality. Item scale ranges from minimum to maximum score of 1-5 for each item, with a higher score indicating a better outcome.
  Intervention process from baseline to follow-up was analyzed using a general linear mixed model, using the item "How often does he/she praise you for doing well?" Time since first baseline clinic visit was computed and analyzed using a mixed model with time, arm, and the time-arm interaction term. The outcome measure data are reported as slopes by arm.
  *NOTE: Intervention process measures were administered biweekly, and we are reporting the calculated mean change per day with 95% confidence intervals.
Time Frame: 3-4 months after baseline (follow-up timepoint)
Measure: Mean (95% Confidence Interval); unit: scores per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 55 | 25
scores per day | .0012 [-.0013 to .0037] | .0045 [.0007 to .0083]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored between baseline (at time of enrollment) to follow-up (generally 3-4 months after enrollment).
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/25
Other Adverse Events (participants affected / at risk) | 0/55 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT02877680/Prot_SAP_000.pdf